CLINICAL TRIAL: NCT05016154
Title: A Randomised Controlled Trial of Online Group CBT for Symptoms of Depression and Anxiety Among University Students in South Africa
Brief Title: Online Psychological Group Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Stellenbosch (Other)
Collaborators: Harvard University (Other); West Virginia University (Other)
Responsible Party: Principal Investigator, Jason Bantjes, Professor, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12977; IRPSD-1681 (Other: Stellenbosch University)
Record Dates: First submitted 2021-08-04; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Depression; Anxiety
Keywords: online group psychological intervention; depression; anxiety; online group Cognitive Behavioural Therapy; App-based interventions; Randomized controlled trial
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Online group CBT intervention (Experimental): Online group CBT delivered via Microsoft Teams (a secure web-based video conferencing platform) in 10 weekly workshops of 60-75 minutes.
  Interventions: Behavioral: Online Group CBT intervention
- SilverCloud guided (Active Comparator): The SilverCloud app is a set of programs and courses that can be completed on a phone, tablet or computer. Students are also contacted by the SilverCloud support team which offers them guidance and support while using the app.
  Silvercloud uses principles borrowed from both a popular type of counseling called Cognitive Behavioral Therapy (CBT) and Mindfulness. Each module takes approximately 40minutes to complete. Students are encouraged to complete at least one module per week.
  Interventions: Behavioral: SilverCloud guided
- SilverCloud unguided (Active Comparator): The SilverCloud app is a set of programs and courses that can be completed on a phone, tablet or computer. Students are encouraged to use the app as they see fit, although guidelines to using the app are provided.
  Silvercloud uses principles borrowed from both a popular type of counseling called Cognitive Behavioral Therapy (CBT) and Mindfulness. Each module takes approximately 40minutes to complete. Students are encouraged to complete at least one module per week.
  Interventions: Behavioral: SilverCloud Unguided
- Mood Flow (Active Comparator): The Moodflow app is a mood tracker and journal that helps students figure out what changes their mood. Students are encouraged to use the app as they see fit, although guidelines to using the app are provided.
  Interventions: Behavioral: Mood Flow

INTERVENTIONS:
Behavioral: Online Group CBT intervention — Group of participants complete 10 weeks of Online Group CBT intervention
  Arms: Online group CBT intervention
Behavioral: SilverCloud guided — Group of participants make use of the SilverCloud guided app
  Arms: SilverCloud guided
Behavioral: SilverCloud Unguided — Group of participants make use of the SilverCloud Unguided app
  Arms: SilverCloud unguided
Behavioral: Mood Flow — Group of participants make use of the Mood Flow app
  Arms: Mood Flow

SUMMARY:
The aim is to assess the effectiveness of online group CBT for reducing symptoms of depression and anxiety among university students. The investigators will conduct a four-arm randomised control trial comparing a 10-session online group CBT intervention to three mental health apps (namely SilverCloud guided, SilverCloud unguided, and Mood Flow).

DETAILED DESCRIPTION:
Email invitations and information about the study will be sent to random samples of students inviting those with symptoms of depression, anxiety, or stress to join the trial.

Students who express interest will be asked to complete an online consent form (providing more detailed information about the study and explaining potential risks and benefits of participation), following which they will complete a baseline assessment. Students who meet inclusion criteria will then be randomly allocated to one of four interventions. Follow-up assessments will be done at 3-, 6- and 12-months post intervention.

The baseline assessment will include measures of depression and anxiety, as well as factors that could potentially predict treatment responses (such as gender, age, substance use, self-harm, adverse childhood experiences, and physical health). Follow-up assessments will include measures of depression and anxiety, as well as substance use, self-harm, and treatment seeking.

The primary outcomes will be symptoms of depression and anxiety as measured by the GAD-7 and PHQ-9.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or older years.
2. Enrolled as a student at Stellenbosch University.
3. Provide Informed Consent.
4. Access to internet to join the online group.

Exclusion Criteria:

1. No internet availability.
2. Did not provide Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline scores in the mean symptoms of depression as measured by the PHQ-9 at 3-months. | Baseline and 3-month follow up assessment for experiment and control interventions groups.
  Determine if a 10-week online group CBT (GCBT) intervention effectively reduces mean scores of depression, between baseline and 3-month follow up, among university students when compared with three control group interventions (i.e., Mood Flow, SilverCloud guided, and SilverCloud unguided).
Change from baseline scores in the mean symptoms of anxiety as measured by the GAD-7 at 3-months. | Baseline and 3-month follow up assessment for experiment and control interventions groups.
  Determine if a 10-week online group CBT (GCBT) intervention effectively reduces mean scores of anxiety, between baseline and 3-month follow up, among university students when compared with three control group interventions (i.e., Mood Flow, SilverCloud guided, and SilverCloud unguided).

CONTACTS AND LOCATIONS:
Overall Officials: Jason Bantjes, PhD, Principal Investigator — University of Stellenbosch
Locations (1):
- Stellenbosch University, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bantjes J, Kazdin AE, Cuijpers P, Breet E, Dunn-Coetzee M, Davids C, Stein DJ, Kessler RC. A Web-Based Group Cognitive Behavioral Therapy Intervention for Symptoms of Anxiety and Depression Among University Students: Open-Label, Pragmatic Trial. JMIR Ment Health. 2021 May 27;8(5):e27400. doi: 10.2196/27400. PMID 34042598

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT05016154/Prot_SAP_000.pdf